CLINICAL TRIAL: NCT02738047
Title: Pharmacogenomic Test Assessment for Medication Management in the Advancement of Medicine
Brief Title: Reduction of Adverse Drug Events and Readmissions
Acronym: RADAR-PGX
Status: Recruiting | Type: Observational
Sponsor: ClinLogic LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 10202016
Record Dates: First submitted 2016-03-28; First posted 2016-04-14 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2023-12

CONDITIONS: Pharmacogenomic Testing for Medication Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 120 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pharmocogenomic test assessment in the medication regimen and disease management for patients under drugs known with genetic variation.

DETAILED DESCRIPTION:
Pharmocogenomic. A multicenter, observational study to evaluate the use of a Pharmocogenomic test assessment in the medication regimen and disease management for patients under drugs known to be influenced by genetic variation.

ELIGIBILITY:
INCLUSION CRITERIA

Patients may be included in the Study if they meet all of the following inclusion criteria:

1. Male or female patients of 25 years of age or older who are able to give their written Informed Consent to participate in a Clinical Study based on voluntary agreement with a thorough explanation of the patient's participation will be provided to them.
2. Patient underwent PGx testing for alleles appropriate to the target drugs within the prior 120 days ("index PGx test assessment");
3. Patient was receiving at least one medication known to be associated with allelic variation at the time of the ("index PGx test assessment"), including over-the- counter medications;
4. Patient has a history of at least one TDAE over the 24-month period preceding the PGx test assessment, or has experienced inadequate efficacy from a target drug.

EXCLUSION CRITERIA

Patients will be excluded from the Study if any of the following criteria apply:

1. Patient is currently hospitalized;
2. Patient's medical and medication history is unavailable over the 120-day period preceding the PGx test assessment;
3. Patient is unable to provide an accurate history due to mental Incapacity;
4. Patient is known to have undergone prior PGx testing for genes specific to the target drug(s), exclusive of the PGx test relating to this Study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are under treatment with several drugs with any of the sequences of biochemical reactions, catalyzed by enzymes, known to be influenced by genetic variation in a patient population.
Sampling Method: Non-Probability Sample
Enrollment: 280000 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Radar, Pharmocogenomic | The period of enrollment is anticipated to be 36 months with a 120- day follow-up period, for total study duration of approximately 40 months from first patient enrolled to completion of follow-up on the last patient in.
  The primary endpoint of the study is the binary occurrence of meaningful change in drug regimen, defined in each patient when:
  1. A genotype known to affect a drug the patient is taking is identified, *and*
  2. The patient's treating physician makes at least one target drug regimen change, dose, substitution, or discontinuation.
  Change in drug dose, substitution, or discontinuation among patients with an identified genotype known to affect a drug the patient is taking as directed. This will be assessed by a quantitative survey.

CONTACTS AND LOCATIONS:
Overall Officials: Haleh Farzanmehr, MD, Principal Investigator — GXL; Haleh Farzanmehr, MD, Study Director — GXL
Locations (1):
- MD@Home, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided